CLINICAL TRIAL: NCT01733680
Title: Amiloride Hydrochloride as an Effective Treatment for ADHD
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study stopped due to lack of recruitment
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 320969
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-10

CONDITIONS: ADHD
Keywords: ADHD; executive function; emotional self-regulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Emotional Regulation | interventions — Amiloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiloride (Active Comparator): Drug: Subjects will take 5mg qd Amiloride for 2 weeks, 10mg qd Amiloride for 3 weeks, 15 mg qd Amiloride for 3 weeks.
  Behavioral: Each week subjects will complete the AISRS, BRIEF-A, and CGI.
  Interventions: Drug: amiloride; Behavioral: Behavioral
- Placebo (Placebo Comparator): Drug: Subjects will take placebo for 8 weeks Behavioral: Each week subjects will complete questionnaires: AISRS, BRIEF-A, and CGI
  Interventions: Behavioral: Behavioral

INTERVENTIONS:
Drug: amiloride — Subjects will take either amiloride hydrochloride or placebo for 8 weeks.
  Arms: Amiloride
Behavioral: Behavioral — Each week of the study, subjects will complete the AISRS, BRIEF-A, and CGI to measure symptom improvement
  Other Names: ADHD symptoms, executive function, emotional self-regulation

SUMMARY:
The investigators are proposing to test a medication derived from our prior studies of the gene SLC9A9. This one gene makes NHE proteins that control how we learn and remember items, which is impaired in ADHD and may cause an inability to plan, prioritize, self-monitor,inhibit, initiate, self-correct, or control one's behavior. The investigators now propose to investigate the therapeutic utility of an NHE inhibitor, amiloride hydrochloride, for the treatment of attention deficit hyperactivity disorder (ADHD) in medication-naïve adults with ADHD.

DETAILED DESCRIPTION:
Our specific aims and hypotheses are as follows:

Primary Aim: Assess the efficacy and adverse effects of amiloride in medication naive ADHD adults in a placebo controlled study. Hypothesis 1: Amiloride will reduce scores on our primary outcome measure, the Adult Attention-Deficit/Hyperactivity Disorder Investigator Symptom Rating Scale (AISRS) and on our secondary outcome, the ADHD specific Clinical Global Impressions (CGI) improvement scale. Hypothesis 2: Amiloride will be well tolerated and will have few side effects in adults with ADHD.

Exploratory Aim 2: Assess effects of amiloride on ADHD-associated clinical features. We will also assess, in an exploratory manner, the effect of amiloride on two clinical features that are not well treated by current ADHD medications: deficits in emotional self-regulation (DESR) and executive function deficit (EFD). Hypothesis 3 predicts that amiloride treatment will reduce symptoms of DESR and of EFD.

We will recruit 40 adults who are diagnosed with ADHD in a double blind placebo controlled study. 20 subjects will receive amiloride hydrochloride and 20 subjects will receive placebo for 8 weeks. Participation in the study requires subjects to meet with the physician for a screening visit, baseline visit and 8 additional weekly visits.

ELIGIBILITY:
Inclusion Criteria:

1. Medication naïve male or female adults ages 18-55 years.
2. A diagnosis of DSM-IV ADHD combined type based on clinical assessment by the study psychiatrist using the Conners Adult ADHD Diagnostic Interview;
3. proficiency in English;
4. A baseline score of 24 or more on the AISRS;
5. ability to swallow pills;
6. ability to report reliably, understand the nature of the study and sign an informed consent document as determined by the study psychiatrist

Exclusion Criteria:

We will exclude potential participants who:

1. have had pharmacologic treatment for ADHD in the past year;
2. are pregnant or nursing;
3. are Investigators or their immediate family (spouse, parent, child, grandparent, or grandchild);
4. have any serious, unstable medical illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease;
5. have severe allergies or multiple adverse drug reactions;
6. have a current or past history of seizures;
7. meet current DSM-IV criteria for anxiety or depression or illicit substance abuse in prior six months (these exclusions are feasible because, although the lifetime comorbidity of ADHD with these disorders is high, we and others have shown that the presence of these disorders at the time of ascertainment for adult ADHD studies is less than 10%);
8. are judged by the study psychiatrist to be at serious suicidal risk.
9. have current or past diagnoses of schizophrenia or bipolar disorder;
10. have a history of hypersensitivity to amiloride or drug class members;
11. have a history of hyperkalemia, diabetes mellitus, renal disease or anuria;
12. have renal impairment Cr > 1.5; or
13. are taking potassium supplements, aldosterone antagonists, tacrolimus or ACE inhibitors.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen V Faraone, PhD, Principal Investigator — SUNY Upstate Medical Unversity; Prashant Kaul, MD, Principal Investigator — VA Medical Center at Syracuse
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via a medical clinic and outside advertisement. Due to the stringent inclusion/exclusion criteria, we were only able to recruit 3 subjects and the physician who was conducting the study chose not to continue and we were unable to find another physician.
Groups:
- Amiloride: Drug: Subjects will take 5mg qd Amiloride for 2 weeks, 10mg qd Amiloride for 3 weeks, 15 mg qd Amiloride for 3 weeks.
  Behavioral: Each week subjects will complete the AISRS, BRIEF-A, and CGI.
  amiloride: Subjects will take either amiloride hydrochloride or placebo for 8 weeks.
  Behavioral: Each week of the study, subjects will complete the AISRS, BRIEF-A, and CGI to measure symptom improvement
Period: Overall Study
Arm/Group | Amiloride | Placebo
Started | 2 | 1
Completed | 2 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1-Amiloride: Subjects received amiloride hydrochloride (5 mg for 2 weeks, 10 mg for 3 week, and 15 mg for 3 weeks.
- Arm 2-Placebo: Subjects received placebo for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm 1-Amiloride | Arm 2-Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3
CGI [Mean (Full Range); unit: units on a scale] — Clinical Global Impressions (CGI)
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
  units on a scale | 4.0 [4.0 to 4.0] | 5 [5 to 5] | 4.33 [4 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Improvement in CGI
Description: CGI Improvement scale: 1=very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse
Time Frame: 8 weeks
Population: There was no statistical analysis done due to the small number of participants in the study
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Amiloride | Placebo
Number analyzed (Participants) | 2 | 1
Units on a scale
  CGI Week 3 | 4 [4 to 4] | 5 [5 to 5]
  CGI Week 4 | 4 [4 to 4] | 3 [3 to 3]
  CGI Week 5 | 4 [4 to 4] | 5 [5 to 5]
  CGI Week 6 | 3.5 [3 to 4] | 5 [5 to 5]
  CGI Week 7 | 4 [4 to 4] | 5 [5 to 5]
  CGI Week 8 | 3.5 [3 to 4] | 5 [5 to 5]
  CGI Week 9 | 3.5 [3 to 4] | 5 [5 to 5]
  CGI Week 10 | 3.5 [3 to 4] | 5 [5 to 5]

2. Secondary Outcome: AISRS, Adult ADHD Investigator Rating Scale
Description: An 18 item clinician administered questionnaire to evaluate ADHD in adults. Responses to questions were 0-None, 1-Mild, 2-Moderate, 3-Severe. A decrease of 30% in the total score would be considered improvement. Total score range is 0-54. A lower score indicates improvement in symptoms. A score of 24 or more indicates symptomatic ADHD.
Time Frame: 8 weeks
Population: Statistical analysis of the outcome data was not done due to the small N.
Measure: Mean (Full Range); unit: Total score
Groups:
- Arm 1-Amiloride: Amiloride was administered for 8 weeks. 5 mg for 2 weeks, 10 mg for 3 weeks and 15 mg for 3 weeks
- Arm 2-Placebo: Subjects were given placebo for 8 weeks
Arm/Group | Arm 1-Amiloride | Arm 2-Placebo
Number analyzed (Participants) | 2 | 1
Total score
  Week 3 | 39 [30 to 48] | 54 [54 to 54]
  Week 4 | 38.5 [29 to 48] | 51 [51 to 51]
  Week 5 | 32.5 [18 to 47] | 50 [50 to 50]
  Week 6 | 31 [20 to 42] | 50 [50 to 50]
  Week 7 | 31 [17 to 45] | 50 [50 to 50]
  Week 8 | 34 [19 to 49] | 50 [50 to 50]
  Week 9 | 26 [14 to 38] | 50 [50 to 50]
  Week 10 | 32.5 [20 to 45] | 50 [50 to 50]

3. Secondary Outcome: The Behavior Rating Inventory of Executive Function-Adult (BRIEF-A)
Description: BRIEF-A is a 75 item self report questionnaire that measures behavior and executive function. For each item the subject is asked "during the past month, how often has each of the following behaviors been a problem?:" The choices are N (never), S (sometimes), O (Often). Total score for the Global Executive Composite used. Raw data were transformed into t-scores, which are standardized scores that indicate the number of standard deviations away from the mean. A T-score of 50 is equal to the mean. Values less than 65 indicate executive function is not a problem and values greater than 65 indicate executive function is often a problem.
Time Frame: 8 weeks
Population: Statistical analysis of the outcome data was not done due to the small N of each group
Measure: Mean (90% Confidence Interval); unit: Global Executive Composite T Score
Groups:
- Arm 1-Amiloride: Subjects received amiloride hydrochloride for 8 weeks. 5 mg/day for 2 weeks, 10 mg/day for 3 weeks, and 15 mg/day for 3 weeks.
Arm/Group | Arm 1-Amiloride | Arm 2-Placebo
Number analyzed (Participants) | 2 | 1
Global Executive Composite T Score
  Week 3 | 66.5 [63.5 to 69.5] | 95 [92 to 98]
  Week 4 | 70.5 [67.5 to 73.5] | 92 [89 to 95]
  Week 5 | 68 [65 to 71] | 96 [93 to 99]
  Week 6 | 68.5 [65.5 to 71.5] | 96 [93 to 99]
  Week 7 | 62.5 [59.5 to 65.5] | 96 [93 to 99]
  Week 8 | 62.5 [59.5 to 65.5] | 96 [93 to 99]
  Week 9 | 62.5 [59.5 to 65.5] | 96 [93 to 99]
  Week 10 | 62 [59 to 65] | 96 [93 to 99]

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Adverse events that were monitored was blood pressure, weight, heart rate, EKG, CBC, TSH, lipid profile, BMP, general malaise, tiredness, headache.
Arm/Group | Amiloride | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

LIMITATIONS AND CAVEATS:
Because of the low number of subjects enrolled in the study, no outcome measures were statistically analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes